CLINICAL TRIAL: NCT02912975
Title: A Randomized Controlled Clinical Trial of Mirror Treatment in the Management of Phantom and Residual Limb Pain in Patients With Trans-tibial Land Mine Amputations in Cambodia
Brief Title: A Clinical Trial of Mirror Treatment for Phantom Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trauma Care Foundation, Norway (Other)
Collaborators: University Hospital of North Norway (Other); NCHADS - Ministry of Health of Cambodia (Other)
Responsible Party: Principal Investigator, Hans Husum, Clinic head, Trauma Care Foundation, Norway
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 975 905 055
Record Dates: First submitted 2016-01-03; First posted 2016-09-23 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Phantom Limb Pain; Complex Regional Pain Syndromes
MeSH Terms: conditions — Phantom Limb; Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirror treatment (Experimental): Five minutes treatment period twice a day for three weeks
  Interventions: Other: Tactile treatment
- Tactile treatment (Active Comparator): Tactile massage twice a day for three weeks
  Interventions: Other: Mirror treatment

INTERVENTIONS:
Other: Mirror treatment — The mirror treatment: The patient sits on a chair, both knees in 90 degrees flexion, both lower limbs undressed, and places a mirror of 100 cm x 25 cm along the trans-tibial amputation stump so that the uninjured limb is reflected in the mirror while the amputation stump can not be seen by the patient. The patient then performs slow repeated movements of the foot from neutral position into maximum flexion while closely observing the reflected image of the uninjured limb - the illusion of a limb regained - in the mirror. The procedure goes on uninterrupted for five minutes in the morning and in the evening in the home of the study patient.
  Arms: Tactile treatment
Other: Tactile treatment — In Tactile Treatment five different sensory stimuli is applied repeatedly to the skin of the affected part of the limb, in the actual case to the amputated limb from ten cm above the knee joint and distally to include the entire amputation stump: gentle touch with a feather, a brush, a piece of paper, a stone and a wooden stick. The stimuli are applied two times daily for five 5 minutes each time, one minute per material.
  Arms: Mirror treatment

SUMMARY:
A randomized controlled clinical to examine the effect of mirror therapy on phantom pain and residual limb pain in patients with traumatic transtibial amputations in Cambodia. The study will be conducted with a semi-crossover design using self-rated pain and function as the main result variables.

DETAILED DESCRIPTION:
The study will be conducted in two phases: Firstly, the effects of mirror treatment (M) versus tactile treatment (T) will be compared in an open, randomized, semi-cross-over case-control design study. The second phase includes the responders from the initial treatment (M or T), the duration of the initial treatment effect will be observed, and the effect of a second round of similar treatment will be registered.

Phase one: The study patients will be randomized for M or T treatment. The main outcome variables will be gathered before the initial randomization and after an initial treatment period of three weeks. Non-responders (NR) will be allocated for an immediate second three-weeks treatment period of combined treatment (M+T); the responders (R) of the M, T and M+T enter the second phase of the study. The M+T non-responders discontinue the study.

Phase two: The responders will be observed for a period of maximum three months. When symptoms of phantom limb pain and/or CRPS resume, the patients will undergo a second treatment period with the same treatment as during phase one. The duration of the second treatment period will be maximum three weeks, but each patient may decide to interrupt the treatment at an earlier stage if he finds the effect satisfactory. The main outcome indicators will be gathered at the start and the end of the second treatment period.

The study closes at the end of the second treatment period. For both study phases the treatment effects will be compared between the strata and also inside each stratum, using each patient as his own control.

ELIGIBILITY:
Inclusion Criteria:

* Present age >16 years.
* Unilateral trans-tibial land mine amputation more than 12 months before entering the study.
* Suffering from phantom limb pain and/or CRPS-2.

Exclusion Criteria:

* Amputation stump anomalies that require surgical reconstructions such as chronic infections, neuroma or major soft tissue deformities.
* Chronic alcoholism or drug abuse.
* Loss or deformities of limbs other than the actual amputation.
* Mental and/or cognitive disorders making self-reporting unreliable.

Min Age: 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain | Change after three months as compared to preintervention level
  Assessed by self-rating by each study patient

OTHER OUTCOMES:
Physical function | Change after three months as compared to preintervention level
  Assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Snorre Sollied, MD, PhD, Study Director — Department of Intensive Care, University Hospital North Norway
Locations (1):
- Trauma Care Foundation Cambodia, Battambang, Cambodia